CLINICAL TRIAL: NCT02463747
Title: Prospective Unblinded Randomized Trial to Examine Short vs Prolonged Antibiotic Treatment for Hospitalized Hemato-oncology Patients With Febrile Neutropenia
Brief Title: Short vs Prolonged Antibiotic Treatment for Hospitalized Hemato-oncology Patients With Febrile Neutropenia
Acronym: RR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director of R & D - Tel Aviv Sourasky M C, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0143-15-TLV
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Fever; Febrile Neutropenia
Keywords: Neutropenic fever; extended infusion; beta-lactam; empiric antibiotic treatment
MeSH Terms: conditions — Fever; Febrile Neutropenia | interventions — Piperacillin, Tazobactam Drug Combination; Ceftazidime; Meropenem; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Infusion of antibiotics (Experimental): Prolonged (4 hours) Infusion of antibiotics.
  Intervention:
  Primary care would be one of three options:
  1. Piperacillin/tazobactam : 4.5gr, TID, I.V.
     Or
  2. Fortum (Ceftazidim): 2.0gr, TID, I.V. - for penicillin-sensitive patients.
     Or
  3. Meropenem: 1.0gr, TID, I.V.
  Supplementation of Vancomycin will be at the discretion of the treating physician.
  Interventions: Drug: Piperacillin/tazobactam; Drug: Ceftazidim; Drug: Meropenem; Drug: Vancomycin
- Fixed time infusion of antibiotics (Active Comparator): Fixed time (half and hour) infusion of antibiotics.
  Intervention:
  Primary care would be one of three options:
  1. Piperacillin/tazobactam : 4.5gr, TID, I.V.
     Or
  2. Fortum (Ceftazidim): 2.0gr, TID, I.V. - for penicillin-sensitive patients.
     Or
  3. Meropenem: 1.0gr, TID, I.V.
  Supplementation of Vancomycin will be at the discretion of the treating physician/
  Interventions: Drug: Piperacillin/tazobactam; Drug: Ceftazidim; Drug: Meropenem; Drug: Vancomycin

INTERVENTIONS:
Drug: Piperacillin/tazobactam — Initial treatment will be with Piperacillin + Tazobactam
  Other Names: Tazocin
Drug: Ceftazidim — Patient with sensitivity to penicillin will receive Ceftazidim
  Other Names: Fortum
Drug: Meropenem — In cases of hypotension that do not respond to fluids resuscitation , and in consultation with the infectious diseases unit - we will start empirical treatment with Meropenem
  Other Names: Ceftazidim
Drug: Vancomycin — Supplementation of Vancomycin will be at the discretion of the treating physician
  Other Names: Non

SUMMARY:
Neutropenic fever is a life threatening condition that is not rare in patients suffering from hematologic disorders, and of paramount importance to early and effective treatment. In this trial we concentrate on hospitalized patients with hematologic malignancies who develop neutropenic fever.

In recent years, several studies were conducted to examine possible changes in the conventional empirical treatment, assuming that administration of the antibiotics in a prolonged infusion would allow for a greater fT > MIC that will lead to a better efficacy.

These studies were carried out in different populations and there is only limited information about the importance of continuous infusion therapy in patients with hematologic diseases with neutropenic fever.

Research goals: The main goal is to compare between two groups of hematologic patients with neutropenic fever, The first group will receive antibiotic therapy in extended infusion, and the second (control) group will receive the treatment in a fixed time.

DETAILED DESCRIPTION:
METHODS: Each patient who will be hospitalized in the Department of Bone Marrow Transplantation and which meets the Inclusion criteria for, will be offered to participate in the study. If fever appears during hospitalization empirical treatment of neutropenia will be initiated performed in accordance with the allocation of the patient in the study. Therapeutic success is defined as a combination of several clinical parameters, including: a decline in Fever, the recurrence of fever and improvement in infection.

METHODS: Study format - Prospective unblinded randomized trial.

Neutropenic fever measurement will be set above the fold of 38.3 ° C or fever over 38.0 ° C lasting more than an hour. Neutropenia is defined as absolute neutrophil count (ANC) less than 500 cells / mm3, or expected to fall below this value for the next 48 hours.

Primary care would be one of three options:

1. Tazocin: 4.5gr, TID, I.V. Or
2. Fortum (Ceftazidim): 2.0gr, TID, I.V. - for penicillin-sensitive patients. Or
3. Meropenem: 1.0gr, TID, I.V. - In cases of hypotension not responding to fluids resuscitation, and in consultation with the infectious diseases unit - we will start empirical treatment with Meropenem.

Supplementation of Vancomycin will be at the discretion of the treating physician.

Antibiotic therapy will be replaced, in coordination with the Department of Infectious Diseases in the following cases:

1. The fever does not decrease after 24 hours
2. The patient is not hemodynamically stable or developes an organ failure
3. Evolving of sensitivity response (allergy) suspected to be a response to antibiotic patient is treated with.
4. sensitivity response was received from the laboratory culture Bacteriologist demanding a change in antibiotics.

Replacement of antibiotic therapy is defined as a failure as defined by the primary endpoint. In such a case, continued treatment of the patient would be according to the BMT unit protocol for treatment for neutropenic fever.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to sign an informed consent form
2. Hospitalized patients for one of the following reasons:

   * Induction or consolidation for Acute Leukemia
   * Patients Hospitalized for Autologous BMT
   * Patients Hospitalized for Allogeneic BMT.

Exclusion Criteria:

1. Patients under the age of 18.
2. Patients who are unable to provide informed consent.
3. Patients with acute lymphatic leukemia hospitalized for maintenance treatment
4. Patients who will not be staying for the entire duration of neutropenia in house.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
A successful response to treatment | Interim analysis is planed after 1 year , when a recruitment of 50 patients is expected
  A successful response to treatment will be defined by a combination of all the following:
  A. A defervescence of fever for at least 48 hours. B. Disappearance or improvement of clinical signs and symptoms of infection.
  C. No: bacteremia / re-emergence of fever / signs of infection within 5 days from starting of treatment.

SECONDARY OUTCOMES:
Breakthrough fever or Additional bacteremia | 5 days after primary treatment
Clostridium difficile infection | For the duration of hospital stay - an expected average of 4 weeks
Survival | During 30 days from begining of treatment
Duration of Hospitalization | For the duration of hospital stay - an expected average of 4 weeks
Number of days of Neutropenia | For the duration of hospital stay - an expected average of 4 weeks
Any systemic organ Failure (Renal / Hepatic / Cardio or pulmonary) | For the duration of hospital stay - an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ron Ram, MD, Principal Investigator — Head of BMt Unit / hematology division
Locations (1):
- Tel-Aviv Sourasky Medicak center / BMT Unit, Tel Aviv, Israel

REFERENCES:
- [Derived] Ram R, Halavy Y, Amit O, Paran Y, Katchman E, Yachini B, Kor S, Avivi I, Ben-Ami R. Extended vs Bolus Infusion of Broad-Spectrum beta-Lactams for Febrile Neutropenia: An Unblinded, Randomized Trial. Clin Infect Dis. 2018 Sep 28;67(8):1153-1160. doi: 10.1093/cid/ciy258. PMID 29608680